**STUDY TITLE:** Evaluating a Digital Intervention for Binge Eating and Weight Management among Adults with Food Insecurity

NCT NUMBER: NCT06348251

**DATE:** November 15, 2025

## **Statistical Analysis Plan**

Feasibility of study procedures is based on study recruitment rates and study retention rates. Metrics of feasibility will be calculated using descriptives (i.e., means and standard deviations).